CLINICAL TRIAL: NCT02081014
Title: A Randomized, Phase 2a, Blinded, 3-Way Crossover Dose-Ranging Study With G-Pen Mini™ (Glucagon Injection) to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics in Patients With Type 1 Diabetes Mellitus (T1DM)
Brief Title: Safety and Efficacy Study of Mini-Dose Glucagon (G-Pen Mini) in Patients With Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xeris Pharmaceuticals (Industry)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Emissary International LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: XSMP-201; 1R44DK096715-01A1 (NIH)
Record Dates: First submitted 2014-03-04; First posted 2014-03-07 (Estimated); Results first posted 2016-05-16 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-03

CONDITIONS: Hypoglycemia
Keywords: Hypoglycemia; Glucagon; Diabetes
MeSH Terms: conditions — Hypoglycemia; Diabetes Mellitus | interventions — Glucagon

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- G-Pen Mini™ (glucagon injection) 75 ug (Experimental): G-Pen Mini™ (glucagon injection), two 75 microgram subcutaneous injections given approximately 4-5 hours apart
  Interventions: Drug: G-Pen Mini™ (glucagon injection)
- G-Pen Mini™ (glucagon injection) 150 ug (Experimental): G-Pen Mini™ (glucagon injection), two 150 microgram subcutaneous injections given approximately 4-5 hours apart
  Interventions: Drug: G-Pen Mini™ (glucagon injection)
- G-Pen Mini™ (glucagon injection) 300 ug (Experimental): G-Pen Mini™ (glucagon injection), two 300 microgram subcutaneous injections given approximately 4-5 hours apart
  Interventions: Drug: G-Pen Mini™ (glucagon injection)

INTERVENTIONS:
Drug: G-Pen Mini™ (glucagon injection) — stable, pre-mixed, liquid glucagon for subcutaneous injection
  Other Names: mini-dose glucagon

SUMMARY:
The purpose of the study is to demonstrate that mini-doses of stable liquid glucagon (G-Pen Mini) produced by Xeris Pharmaceuticals are safe and effective as a treatment for mild to moderate hypoglycemia, a complication of diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects on insulin infusion pump therapy for treatment of type 1 diabetes
2. Between the ages of 18 and 50 years of age, inclusive, at Screening.
3. Females of childbearing potential with a negative serum pregnancy test prior at screening and negative urine pregnancy tests prior to the Treatment visits, using an approved forms of contraception for the duration of participation in the study (i.e. until after last dose).
4. Male subjects are required to use a condom and another of the methods of contraception in #3 above starting at Randomization and for the duration of the study.
5. Hemoglobin A1c (HbA1c) < 9.0 %.
6. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
7. Subjects must be willing and able to comply with scheduled visits, treatment, laboratory tests and study procedures.

Exclusion Criteria:

1. Clinical evidence of microvascular complication(s) other than mild microalbuminuria or history of mild non-proliferative retinopathy
2. Any chronic diseases or illness that interferes with glucose metabolism, except for T1DM, or medications other than hypothyroidism on appropriate thyroid hormone replacement.
3. Blood pressure (BP) readings at Screening where Systemic BP <90 or >140 mm Hg, and Diastolic BP <50 or >90 mm Hg.
4. Cardiovascular event within 6 months prior to screening such as unstable angina, acute coronary syndrome, myocardial infarction, therapeutic coronary procedure (e.g., stent placement, Percutaneous Transluminal Coronary Angioplasty (PTCA), Coronary Artery By-pass Grafting (CABG)), stroke or transient ischemic attack.
5. Study participants who are pregnant at Screening.
6. Breast feeding must be discontinued if a subject wishes to participate in this study.
7. Positive test for hepatitis B, hepatitis C, or HIV found at Screening.
8. Positive urine drug test for illicit drugs at Screening.
9. History of allergies to glucagon, glucagon-like products or to any of the excipients in the investigational formulation.
10. Known presence of hereditary problems of glycogen storage disease, galactose and /or lactose intolerance
11. Administration of glucagon more than once within the three (3) months prior to Screening
12. Subjects with any of the following abnormalities in clinical laboratory tests at Screening, confirmed by a single repeat, if necessary:

    * Hemoglobin (Hb) below the lower limits of normal for the laboratory
    * Total bilirubin above the upper limits of normal for the laboratory
    * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) above the upper limits of normal for the laboratory
    * Creatinine above the upper limits of normal for the laboratory
13. History of regular alcohol consumption as defined by alcohol intake in a quantity exceeding 7 drinks per week for females or 14 drinks per week for males, where 1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor.
14. Participation in other studies involving administration of an investigational drug or device within 30 days or 5 half-lives, whichever is longer, before screening for the current study and during participation in the current study
15. Whole blood donation of 1 pint (500 mL) within 8 weeks prior to Screening. Donations of plasma, packed red blood cells, platelets or quantities less than 500 mL are allowed at investigator discretion.
16. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2014-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Morey W Haymond, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Children's Nutritional Research Center, Texas Children's Hospital, Houston, Texas, United States

REFERENCES:
- [Result] Haymond MW, Redondo MJ, McKay S, Cummins MJ, Newswanger B, Kinzell J, Prestrelski S. Nonaqueous, Mini-Dose Glucagon for Treatment of Mild Hypoglycemia in Adults With Type 1 Diabetes: A Dose-Seeking Study. Diabetes Care. 2016 Mar;39(3):465-8. doi: 10.2337/dc15-2124. Epub 2016 Feb 9. PMID 26861921

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 13 adults < 50 years of age with type 1 diabetes were recruited over a period of 5 months to receive treatment at a university-affiliated state hospital-based endocrinology clinic.
Pre-assignment Details: A total of 13 subjects were randomized to treatment. Due to poor venous access an IV could not be started in one subject, so only 12 subjects received treatment.
Groups:
- G-Pen Mini™ Dose Order: 75, 150 & 300 Micrograms: G-Pen Mini™ (glucagon injection): two 75 microgram (ug) subcutaneous (SC) injections at treatment visit 1, followed by a 2-21 day washout, then two 150 ug SC injections at treatment visit 2, followed by a 2-21 day washout, and finally two 300 ug SC injections at treatment visit 3.
- G-Pen Mini™ Dose Order: 75, 300 & 150 Micrograms: G-Pen Mini™ (glucagon injection): two 75 ug SC injections at treatment visit 1, followed by a 2-21 day washout, then two 300 ug SC injections at treatment visit 2, followed by a 2-21 day washout, and finally two 150 ug SC injections at treatment visit 3.
- G-Pen Mini™ Dose Order: 150, 75 & 300 Micrograms: G-Pen Mini™ (glucagon injection): two 150 ug SC injections at treatment visit 1, followed by a 2-21 day washout, then two 75 ug SC injections at treatment visit 2, followed by a 2-21 day washout, and finally two 300 ug SC injections at treatment visit 3.
- G-Pen Mini™ Dose Order: 150, 300 & 75 Micrograms: G-Pen Mini™ (glucagon injection): two 150 ug SC injections at treatment visit 1, followed by a 2-21 day washout, then two 300 ug SC injections at treatment visit 2, followed by a 2-21 day washout, and finally two 150 ug SC injections at treatment visit 3.
- G-Pen Mini™ Dose Order: 300, 75 & 150 Micrograms: G-Pen Mini™ (glucagon injection): two 300 ug SC injections at treatment visit 1, followed by a 2-21 day washout, then two 75 ug SC injections at treatment visit 2, followed by a 2-21 day washout, and finally two 150 ug SC injections at treatment visit 3.
- G-Pen Mini™ Dose Order: 300, 150 & 75 Micrograms: G-Pen Mini™ (glucagon injection): two 300 ug SC injections at treatment visit 1, followed by a 2-21 day washout, then two 150 ug SC injections at treatment visit 2, followed by a 2-21 day washout, and finally two 75 ug SC injections at treatment visit 3.
Period: Overall Study
Arm/Group | G-Pen Mini™ Dose Order: 75, 150 & 300 Micrograms | G-Pen Mini™ Dose Order: 75, 300 & 150 Micrograms | G-Pen Mini™ Dose Order: 150, 75 & 300 Micrograms | G-Pen Mini™ Dose Order: 150, 300 & 75 Micrograms | G-Pen Mini™ Dose Order: 300, 75 & 150 Micrograms | G-Pen Mini™ Dose Order: 300, 150 & 75 Micrograms
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized subjects who received at least one dose of study drug
Groups:
- Total Study Group: Includes all 12 treated subjects
Arm/Group | Total Study Group
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 11
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.4 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12
HbA1c [Mean (Standard Deviation); unit: percent] | 7.7 (0.48)
Body Weight [Mean (Standard Deviation); unit: kg] | 73.6 (12.08)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 11.6 (6.02)

OUTCOME MEASURES:

1. Primary Outcome: Serious Adverse Events
Description: Number of serious adverse events (SAEs) per treatment
Time Frame: From first dose until follow-up call, up to 7 weeks per subject
Population: All randomized subjects who received at least one dose of study drug
Measure: Number; unit: participants
Arm/Group | G-Pen Mini™ (Glucagon Injection) 75 ug | G-Pen Mini™ (Glucagon Injection) 150 ug | G-Pen Mini™ (Glucagon Injection) 300 ug
Number analyzed (Participants) | 12 | 12 | 12
participants | 0 | 0 | 0

2. Secondary Outcome: Glucagon Cmax (Fasting)
Description: Pharmacokinetic parameter: Maximum concentration of glucagon
Time Frame: Approximately 15 and 0 minutes before each injection and at 5, 10, 15, 20, 30, 45, 60, 120 and 180 minutes post-injection
Population: All randomized subjects who received at least one dose of study drug
Measure: Mean (Standard Error); unit: pg/ml
Groups:
- G-Pen Mini™ (Glucagon Injection) 75 ug: G-Pen Mini™ (glucagon injection), a single 75 microgram subcutaneous injection given to subjects after an overnight fast
- G-Pen Mini™ (Glucagon Injection) 150 ug: G-Pen Mini™ (glucagon injection), a single 150 microgram subcutaneous injection given given to subjects after an overnight fast
- G-Pen Mini™ (Glucagon Injection) 300 ug: G-Pen Mini™ (glucagon injection), a single 300 microgram subcutaneous injection given given to subjects after an overnight fast
Arm/Group | G-Pen Mini™ (Glucagon Injection) 75 ug | G-Pen Mini™ (Glucagon Injection) 150 ug | G-Pen Mini™ (Glucagon Injection) 300 ug
Number analyzed (Participants) | 12 | 12 | 12
pg/ml | 233.8 (34) | 380.7 (34) | 663.6 (34)
Statistical Analysis 1: Comparison: G-Pen Mini™ (Glucagon Injection) 75 ug vs G-Pen Mini™ (Glucagon Injection) 150 ug; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Point estimate ratio = 0.62, Standard Error of Mean 0.07 — Geometric means
Statistical Analysis 2: Comparison: G-Pen Mini™ (Glucagon Injection) 75 ug vs G-Pen Mini™ (Glucagon Injection) 300 ug; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Point estimate ratio = 0.35, Standard Error of Mean 0.04 — Geometric means
Statistical Analysis 3: Comparison: G-Pen Mini™ (Glucagon Injection) 150 ug vs G-Pen Mini™ (Glucagon Injection) 300 ug; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Point estimate ratio = 0.57, Standard Error of Mean 0.06 — Geometric means

3. Secondary Outcome: Glucagon Cmax (Post-insulin)
Description: Pharmacokinetic parameter: Maximum concentration of glucagon
Time Frame: Approximately 15 and 0 minutes before each injection and at 5, 10, 15, 20, 30, 45, 60, and 120 minutes post-injection
Population: All randomized subject who received at least one dose of study drug
Measure: Mean (Standard Error); unit: pg/ml
Groups:
- G-Pen Mini™ (Glucagon Injection) 75 ug: G-Pen Mini™ (glucagon injection), a single 75 microgram subcutaneous injection given to subjects in a state of mild hypoglycemia
- G-Pen Mini™ (Glucagon Injection) 150 ug: G-Pen Mini™ (glucagon injection), a single 150 microgram subcutaneous injection given to subjects in a state of mild hypoglycemia
- G-Pen Mini™ (Glucagon Injection) 300 ug: G-Pen Mini™ (glucagon injection), a single 300 microgram subcutaneous injection given to subjects in a state of mild hypoglycemia
Arm/Group | G-Pen Mini™ (Glucagon Injection) 75 ug | G-Pen Mini™ (Glucagon Injection) 150 ug | G-Pen Mini™ (Glucagon Injection) 300 ug
Number analyzed (Participants) | 12 | 12 | 12
pg/ml | 253.4 (30.1) | 335.4 (30.1) | 561.7 (29.9)
Statistical Analysis 1: Comparison: G-Pen Mini™ (Glucagon Injection) 75 ug vs G-Pen Mini™ (Glucagon Injection) 150 ug; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Point estimate ratio = 0.74, Standard Error of Mean 0.06 — Geometric means
Statistical Analysis 2: Comparison: G-Pen Mini™ (Glucagon Injection) 75 ug vs G-Pen Mini™ (Glucagon Injection) 300 ug; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Point estimate ratio = 0.44, Standard Error of Mean 0.04 — Geometric means
Statistical Analysis 3: Comparison: G-Pen Mini™ (Glucagon Injection) 150 ug vs G-Pen Mini™ (Glucagon Injection) 300 ug; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Point estimate ratio = 0.59, Standard Error of Mean 0.05 — Geometric means

4. Secondary Outcome: Glucagon Area Under the Curve (AUC) (Fasting)
Description: Pharmacokinetic parameter: Area under the glucagon concentration curve from 0 to 120 minutes
Time Frame: Approximately 15 and 0 minutes before each injection and at 5, 10, 15, 20, 30, 45, 60, and 120 minutes post-injection
Population: All randomized subjects who received at least one dose of study drug
Measure: Mean (Standard Error); unit: (pg/ml)*hour
Arm/Group | G-Pen Mini™ (Glucagon Injection) 75 ug | G-Pen Mini™ (Glucagon Injection) 150 ug | G-Pen Mini™ (Glucagon Injection) 300 ug
Number analyzed (Participants) | 12 | 12 | 12
(pg/ml)*hour | 265.4 (35.4) | 389.6 (35.4) | 735.3 (35.4)
Statistical Analysis 1: Comparison: G-Pen Mini™ (Glucagon Injection) 75 ug vs G-Pen Mini™ (Glucagon Injection) 150 ug; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Point point ratio = 0.68, Standard Error of Mean 0.05 — Geometric means
Statistical Analysis 2: Comparison: G-Pen Mini™ (Glucagon Injection) 75 ug vs G-Pen Mini™ (Glucagon Injection) 300 ug; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Point estimate ratio = 0.36, Standard Error of Mean 0.03 — Geometric means
Statistical Analysis 3: Comparison: G-Pen Mini™ (Glucagon Injection) 150 ug vs G-Pen Mini™ (Glucagon Injection) 300 ug; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Point estimate ratio = 0.53, Standard Error of Mean 0.04 — Geometric means

5. Secondary Outcome: Glucagon AUC (Post-insulin)
Description: Pharmacokinetic parameter: Area under the glucagon concentration curve from 0 to 120 minutes
Time Frame: Approximately 15 and 0 minutes before each injection and at 5, 10, 15, 20, 30, 45, 60, and 120 minutes post-injection
Population: All randomized subjects who received at least one dose of study drug
Measure: Mean (Standard Error); unit: (pg/ml)*hour
Arm/Group | G-Pen Mini™ (Glucagon Injection) 75 ug | G-Pen Mini™ (Glucagon Injection) 150 ug | G-Pen Mini™ (Glucagon Injection) 300 ug
Number analyzed (Participants) | 12 | 12 | 12
(pg/ml)*hour | 277.4 (29.9) | 386.8 (29.9) | 635.3 (29.7)
Statistical Analysis 1: Comparison: G-Pen Mini™ (Glucagon Injection) 75 ug vs G-Pen Mini™ (Glucagon Injection) 150 ug; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Point estimate ratio = 0.72, Standard Error of Mean 0.04 — Geometric means
Statistical Analysis 2: Comparison: G-Pen Mini™ (Glucagon Injection) 75 ug vs G-Pen Mini™ (Glucagon Injection) 300 ug; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Point estimate ratio = 0.44, Standard Error of Mean 0.02 — Geometric means
Statistical Analysis 3: Comparison: G-Pen Mini™ (Glucagon Injection) 150 ug vs G-Pen Mini™ (Glucagon Injection) 300 ug; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Point estimate ratio = 0.60, Standard Error of Mean 0.03 — Geometric means

6. Secondary Outcome: Glucagon Tmax (Fasting)
Description: Pharmacokinetic parameter: Time to reach maximum concentration of glucagon
Time Frame: as for outcome 2
Population: All randomized subjects who received at least one dose of study drug
Measure: Mean (Standard Error); unit: minutes
Groups:
- G-Pen Mini™ (Glucagon Injection) 75 ug: G-Pen Mini™ (glucagon injection), a single 75 microgram subcutaneous injection given fo subjects following an overnight fast
- G-Pen Mini™ (Glucagon Injection) 150 ug: G-Pen Mini™ (glucagon injection), a single 150 microgram subcutaneous injection given fo subjects following an overnight fast
- G-Pen Mini™ (Glucagon Injection) 300 ug: G-Pen Mini™ (glucagon injection), a single 300 microgram subcutaneous injection given fo subjects following an overnight fast
Arm/Group | G-Pen Mini™ (Glucagon Injection) 75 ug | G-Pen Mini™ (Glucagon Injection) 150 ug | G-Pen Mini™ (Glucagon Injection) 300 ug
Number analyzed (Participants) | 12 | 12 | 12
minutes | 29.2 (3.6) | 29.8 (3.6) | 36.5 (3.6)
Statistical Analysis 1: Comparison: G-Pen Mini™ (Glucagon Injection) 75 ug vs G-Pen Mini™ (Glucagon Injection) 150 ug; Test type: Superiority or Other; p > 0.05, Mixed Models Analysis; Point esimate ratio = 0.98, Standard Error of Mean 0.14 — Geometric means
Statistical Analysis 2: Comparison: G-Pen Mini™ (Glucagon Injection) 75 ug vs G-Pen Mini™ (Glucagon Injection) 300 ug; Test type: Superiority or Other; p > 0.05, Mixed Models Analysis; Point estimate ratio = 0.78, Standard Error of Mean 0.11 — Geometric means
Statistical Analysis 3: Comparison: G-Pen Mini™ (Glucagon Injection) 150 ug vs G-Pen Mini™ (Glucagon Injection) 300 ug; Test type: Superiority or Other; p > 0.05, Mixed Models Analysis; Point estimate ratio = 0.79, Standard Error of Mean 0.11 — Geometric means

7. Secondary Outcome: Glucagon Tmax (Post-insulin)
Description: Pharmacokinetic parameter: Time to reach maximum concentration of glucagon
Time Frame: Approximately 15 and 0 minutes before each injection and at 5, 10, 15, 20, 30, 45, 60, and 120 minutes post-injection
Population: All randomized subjects who received at least one dose of study drug
Measure: Mean (Standard Error); unit: minutes
Arm/Group | G-Pen Mini™ (Glucagon Injection) 75 ug | G-Pen Mini™ (Glucagon Injection) 150 ug | G-Pen Mini™ (Glucagon Injection) 300 ug
Number analyzed (Participants) | 12 | 12 | 12
minutes | 24 (2.7) | 33.1 (2.7) | 34.1 (2.7)
Statistical Analysis 1: Comparison: G-Pen Mini™ (Glucagon Injection) 75 ug vs G-Pen Mini™ (Glucagon Injection) 150 ug; Test type: Superiority or Other; p > 0.05, Mixed Models Analysis; Point estimate ratio = 0.75, Standard Error of Mean 0.10 — Geometric means
Statistical Analysis 2: Comparison: G-Pen Mini™ (Glucagon Injection) 75 ug vs G-Pen Mini™ (Glucagon Injection) 300 ug; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Point estimate ratio = 0.73, Standard Error of Mean 0.10 — Geometric means
Statistical Analysis 3: Comparison: G-Pen Mini™ (Glucagon Injection) 150 ug vs G-Pen Mini™ (Glucagon Injection) 300 ug; Test type: Superiority or Other; p > 0.05, Mixed Models Analysis; Point estimate ratio = 0.96, Standard Error of Mean 0.13 — Geometric means

8. Secondary Outcome: Glucose Cmax (Fasting)
Description: Pharmacodynamic parameter: Maximum concentration of glucose
Time Frame: as for outcome 2
Population: All randomized subjects who received at least one dose of study drug
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | G-Pen Mini™ (Glucagon Injection) 75 ug | G-Pen Mini™ (Glucagon Injection) 150 ug | G-Pen Mini™ (Glucagon Injection) 300 ug
Number analyzed (Participants) | 12 | 12 | 12
mg/dl | 155.1 (11.2) | 186.2 (11.1) | 213.5 (11.2)
Statistical Analysis 1: Comparison: G-Pen Mini™ (Glucagon Injection) 75 ug vs G-Pen Mini™ (Glucagon Injection) 150 ug; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Point estimate ratio = 0.82, Standard Error of Mean 0.06 — Geometric means
Statistical Analysis 2: Comparison: G-Pen Mini™ (Glucagon Injection) 75 ug vs G-Pen Mini™ (Glucagon Injection) 300 ug; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Point estimate ratio = 0.70, Standard Error of Mean 0.05 — Geometric means
Statistical Analysis 3: Comparison: G-Pen Mini™ (Glucagon Injection) 150 ug vs G-Pen Mini™ (Glucagon Injection) 300 ug; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Point estimate ratio = 0.85, Standard Error of Mean 0.06 — Geometric means

9. Secondary Outcome: Glucose Cmax (Post-insulin)
Description: Pharmacodynamic parameter: Maximum concentration of glucose
Time Frame: Approximately 15 and 0 minutes before each injection and at 5, 10, 15, 20, 30, 45, 60, and 120 minutes post-injection
Population: All randomized subjects who received at least one dose of study drug
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | G-Pen Mini™ (Glucagon Injection) 75 ug | G-Pen Mini™ (Glucagon Injection) 150 ug | G-Pen Mini™ (Glucagon Injection) 300 ug
Number analyzed (Participants) | 12 | 12 | 12
mg/dl | 99.7 (8.6) | 105.7 (8.6) | 122.6 (8.4)
Statistical Analysis 1: Comparison: G-Pen Mini™ (Glucagon Injection) 75 ug vs G-Pen Mini™ (Glucagon Injection) 150 ug; Test type: Superiority or Other; p > 0.05, Mixed Models Analysis; Point estimate ratio = 0.96, Standard Error of Mean 0.08 — Geometric means
Statistical Analysis 2: Comparison: G-Pen Mini™ (Glucagon Injection) 75 ug vs G-Pen Mini™ (Glucagon Injection) 300 ug; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Point estimate ratio = 0.83, Standard Error of Mean 0.06 — Geometric means
Statistical Analysis 3: Comparison: G-Pen Mini™ (Glucagon Injection) 150 ug vs G-Pen Mini™ (Glucagon Injection) 300 ug; Test type: Superiority or Other; p > 0.05, Mixed Models Analysis; Point estimate ratio = 0.86, Standard Error of Mean 0.06 — Geometric means

10. Secondary Outcome: Glucose AUC (Fasting)
Description: Pharmacodynamic parameter: baseline adjusted area under the glucagon concentration curve from 0 to 120 minutes
Time Frame: Approximately 15 and 0 minutes before each injection and at 5, 10, 15, 20, 30, 45, 60, and 120 minutes post-injection
Population: All randomized subjects who received at least one dose of study drug
Measure: Mean (Standard Error); unit: (mg/dl)*minutes
Arm/Group | G-Pen Mini™ (Glucagon Injection) 75 ug | G-Pen Mini™ (Glucagon Injection) 150 ug | G-Pen Mini™ (Glucagon Injection) 300 ug
Number analyzed (Participants) | 12 | 12 | 12
(mg/dl)*minutes | 4872.0 (1495.9) | 8565.2 (1492.8) | 12420.0 (1500.6)
Statistical Analysis 1: Comparison: G-Pen Mini™ (Glucagon Injection) 75 ug vs G-Pen Mini™ (Glucagon Injection) 150 ug; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Mean Difference (Final Values) = -3693.2, Standard Error of Mean 1520.1
Statistical Analysis 2: Comparison: G-Pen Mini™ (Glucagon Injection) 75 ug vs G-Pen Mini™ (Glucagon Injection) 150 ug; Test type: Superiority or Other; p = 0.05, Mixed Models Analysis; Mean Difference (Final Values) = -7548.05, Standard Error of Mean 1542.93
Statistical Analysis 3: Comparison: G-Pen Mini™ (Glucagon Injection) 150 ug vs G-Pen Mini™ (Glucagon Injection) 300 ug; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Mean Difference (Final Values) = -3854.86, Standard Error of Mean 1533.95

11. Secondary Outcome: Glucose AUC (Post-insulin)
Description: Pharmacodynamic parameter: baseline adjusted area under the glucose concentration curve from 0-120 minutes
Time Frame: Approximately 15 and 0 minutes before each injection and at 5, 10, 15, 20, 30, 45, 60, and 120 minutes post-injection
Population: All randomized subjects who received at least one dose of study drug
Measure: Mean (Standard Error); unit: (mg/dl)*minutes
Arm/Group | G-Pen Mini™ (Glucagon Injection) 75 ug | G-Pen Mini™ (Glucagon Injection) 150 ug | G-Pen Mini™ (Glucagon Injection) 300 ug
Number analyzed (Participants) | 12 | 12 | 12
(mg/dl)*minutes | 2263.2 (717.1) | 2408.1 (718.4) | 3928.5 (703.4)
Statistical Analysis 1: Comparison: G-Pen Mini™ (Glucagon Injection) 75 ug vs G-Pen Mini™ (Glucagon Injection) 150 ug; Test type: Superiority or Other; p > 0.05, Mixed Models Analysis; Mean Difference (Final Values) = -144.9, Standard Error of Mean 741.24
Statistical Analysis 2: Comparison: G-Pen Mini™ (Glucagon Injection) 75 ug vs G-Pen Mini™ (Glucagon Injection) 300 ug; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Mean Difference (Final Values) = -1665.32, Standard Error of Mean 696.97
Statistical Analysis 3: Comparison: G-Pen Mini™ (Glucagon Injection) 150 ug vs G-Pen Mini™ (Glucagon Injection) 300 ug; Test type: Superiority or Other; p > 0.05, Mixed Models Analysis; Mean Difference (Final Values) = -1520.39, Standard Error of Mean 700.92

12. Secondary Outcome: Glucose Tmax (Fasting)
Description: Pharmacodynamic parameter: Time to reach maximum concentration of glucose
Time Frame: as for outcome 2
Population: All randomized subjects who received at least one dose of study drug
Measure: Mean (Standard Error); unit: minutes
Arm/Group | G-Pen Mini™ (Glucagon Injection) 75 ug | G-Pen Mini™ (Glucagon Injection) 150 ug | G-Pen Mini™ (Glucagon Injection) 300 ug
Number analyzed (Participants) | 12 | 12 | 12
minutes | 81.5 (10.2) | 80.7 (10.2) | 67.8 (10.3)
Statistical Analysis 1: Comparison: G-Pen Mini™ (Glucagon Injection) 75 ug vs G-Pen Mini™ (Glucagon Injection) 150 ug; Test type: Superiority or Other; p > 0.05, Mixed Models Analysis; Point estimate ratio = 0.41, Standard Error of Mean 0.32 — Geometric means
Statistical Analysis 2: Comparison: G-Pen Mini™ (Glucagon Injection) 75 ug vs G-Pen Mini™ (Glucagon Injection) 300 ug; Test type: Superiority or Other; p > 0.05, Mixed Models Analysis; Point estimate ratio = 0.43, Standard Error of Mean 0.34 — Geometric means
Statistical Analysis 3: Comparison: G-Pen Mini™ (Glucagon Injection) 150 ug vs G-Pen Mini™ (Glucagon Injection) 300 ug; Test type: Superiority or Other; p > 0.05, Mixed Models Analysis; Point estimate ratio = 1.05, Standard Error of Mean 0.81 — Geometric means

13. Secondary Outcome: Glucose Tmax (Post-insulin)
Description: Pharmacodynamic parameter: Time to reach maximum concentration of glucose
Time Frame: Approximately 15 and 0 minutes before each injection and at 5, 10, 15, 20, 30, 45, 60, and 120 minutes post-injection
Population: All randomized subjects who received at least one dose of study drug
Measure: Mean (Standard Error); unit: minutes
Arm/Group | G-Pen Mini™ (Glucagon Injection) 75 ug | G-Pen Mini™ (Glucagon Injection) 150 ug | G-Pen Mini™ (Glucagon Injection) 300 ug
Number analyzed (Participants) | 12 | 12 | 12
minutes | 53.5 (7.1) | 69.5 (7.1) | 57.4 (6.9)
Statistical Analysis 1: Comparison: G-Pen Mini™ (Glucagon Injection) 75 ug vs G-Pen Mini™ (Glucagon Injection) 150 ug; Test type: Superiority or Other; p > 0.05, Mixed Models Analysis; Point estimate ratio = 0.23, Standard Error of Mean 0.29 — Geometric means
Statistical Analysis 2: Comparison: G-Pen Mini™ (Glucagon Injection) 75 ug vs G-Pen Mini™ (Glucagon Injection) 300 ug; Test type: Superiority or Other; p > 0.05, Mixed Models Analysis; Point estimate ratio = 0.73, Standard Error of Mean 0.88 — Geometric means
Statistical Analysis 3: Comparison: G-Pen Mini™ (Glucagon Injection) 150 ug vs G-Pen Mini™ (Glucagon Injection) 300 ug; Test type: Superiority or Other; p > 0.05, Regression, Linear; Point estimate ratio = 3.23, Standard Error of Mean 3.84 — Geometric means

ADVERSE EVENTS:
Arm/Group | G-Pen Mini™ (Glucagon Injection) 75 ug | G-Pen Mini™ (Glucagon Injection) 150 ug | G-Pen Mini™ (Glucagon Injection) 300 ug
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 10/12 | 11/12 | 11/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | G-Pen Mini™ (Glucagon Injection) 75 ug (N=12) | G-Pen Mini™ (Glucagon Injection) 150 ug (N=12) | G-Pen Mini™ (Glucagon Injection) 300 ug (N=12)
blurred vision (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4)
paresthesia (Skin and subcutaneous tissue disorders) | 8 (13) | 8 (13) | 9 (16) — at injection site
hypoesthesia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) — at injection site
nodule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — at injection site
pain (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (4) | 3 (5) — at injection site
bruising (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — at injection site
erythema (Skin and subcutaneous tissue disorders) | 6 (7) | 7 (7) | 6 (7) — at injection site
edema (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (5) | 4 (5) — at injection site
hypoglycemia (Injury, poisoning and procedural complications) | 2 (3) | 2 (2) | 1 (2)
muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
headache (Nervous system disorders) | 1 (2) | 1 (1) | 0 (0)
pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — in fingers
Skin reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — reaction to adhesive used to secure IV line

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No